# Cover page

| Official Title: |
|-------------------------------------------------------------------|
| Incidence of Postoperative Cognitive Decline in Surgical Patients |
| With Preexisting Cognitive Impairment: A Prospective Cohort Study |
| ClinicalTrials.gov Identifier (NCT Number): |
| Document Type: |
| Study Protocol |
| Version Number: |
| No.1 |
| Version Date: |
| May 4, 2025 |
| Principal Investigator: |
| [Yaqian Yu, MN] |
| [Department of Operating room, Peking University Shenzhen |
| Hospital] |
| Sponsor: |

Peking University Shenzhen Hospital

#### **Official Title:**

Incidence of Postoperative Cognitive Decline in Surgical Patients
With Preexisting Cognitive Impairment: A Prospective Cohort Study

## 1. Background

Cognitive impairment is prevalent among the elderly population, with increasing rates as global aging accelerates. Preexisting cognitive impairment (PreCI) in surgical patients is associated with a higher incidence of postoperative cognitive decline (POCD), delirium, hospital readmission, and mortality. However, data regarding the incidence of POCD in Chinese patients with PreCI undergoing elective non-cardiac surgery under general anesthesia is currently lacking. This study aims to fill this evidence gap by prospectively investigating the incidence of POCD in this patient population.

### 2. Objectives

# **Primary Objective:**

To determine the incidence of postoperative cognitive decline (POCD) at 3 months after surgery in elderly patients (≥60 years) with preexisting cognitive impairment undergoing elective non-cardiac surgery under general anesthesia.

### **Secondary Objectives:**

To evaluate the incidence of POCD at 12 months postoperatively.

To assess neuropsychiatric symptoms (NPI-Q), functional abilities (BADL, IADL), and dementia severity (CDR) at 3 and 12 months postoperatively.

# 3. Study Design

A single-center, prospective, single-arm cohort study with a normative comparison group for RCI-based incidence calculation.PreCI Surgical Group: Elderly patients with cognitive impairment undergoing elective general anesthesia non-cardiac surgery. Normative Comparison Group: Cognitively normal elderly subjects for reference data of natural cognitive change over time.

# 4. Study Population

### **Inclusion Criteria (PreCI Group):**

- -Age  $\geq$  60 years
- -Diagnosed as having mild cognitive impairment or mild dementia by MMSE and MoCA-B screening
  - -Scheduled for elective non-cardiac surgery under general anesthesia

#### **Exclusion Criteria:**

- -Expected difficulty in neuropsychological assessment (e.g., severe hearing/visual impairments, language barrier)
  - -Residence outside Shenzhen

## **Normative Comparison Group:**

-Age  $\geq$  60 years

-No history of general anesthesia surgery within the past 12 months

-Mini-Cog score > 1

### **Exclusion Criteria:**

-Planned elective surgery under general anesthesia within the next

12 months

-History of suspected or diagnosed cognitive impairment, or

screening indicating cognitive impairment using MMSE and MoCA-B

-Expected difficulty in completing neuropsychological assessments

(e.g., inability to communicate in Mandarin, blindness, or deafness)

-Usual residence outside Shenzhen

#### 5. Outcome Measures

# **Primary Outcome:**

Incidence of POCD at 3 months postoperatively, defined using the Reliable Change Index (RCI) methodology.

# **Secondary Outcomes:**

Incidence of POCD at 12 months

NPI-Q, BADL, IADL, and CDR scores at 3 and 12 months

#### 6. Assessment Tools

Mini-Cog

**MMSE** 

MoCA-B

NPI-Q

CDR

BADL, IADL

## 7. Sample Size Estimation

PreCI group: 252 patients (accounting for 15% attrition, based on estimated 14.9% POCD incidence at 3 months)

Normative group: 88 participants (allowing for 15% attrition)

# 8. Statistical Analysis Plan (SAP)

### 8.1 Descriptive Analysis:

Continuous variables will be expressed as mean  $\pm$  SD or median (IQR) as appropriate. Categorical variables will be presented as frequencies and percentages.

#### **8.2 Incidence of POCD:**

POCD defined by RCI  $\leq$  -1.96 in at least two cognitive domains or composite Z-score  $\leq$  -1.96.

Frequencies and percentages reported at each follow-up time point.

Subgroup analysis based on surgery type, anesthesia type, baseline cognitive scores.

Intention-to-treat (ITT) analysis applied.

# **8.3 Handling of Missing Data:**

Missing data imputed using multiple imputation techniques.

Sensitivity analyses conducted to evaluate robustness of results.

## 8.4 Adjustment for Confounding:

Multivariable logistic regression used to adjust for potential confounders: age, sex, education, comorbidities, surgery type.

### **8.5 Statistical Software:**

All analyses performed using R software

# 9. Data Management

Data recorded via electronic and paper CRFs. Regular data monitoring, double data entry, and periodic audits to ensure data quality.

### 10. Ethics and Informed Consent

Study approved by the Ethics Committee of Peking University
Shenzhen Hospital. Written informed consent obtained from all
participants or their legal representatives before enrollment.

### 11. Publication Plan

Results will be published in peer-reviewed journals and presented at relevant academic conferences.